CLINICAL TRIAL: NCT01451242
Title: The Reliability of Heart Rate Variability Measurements Among Patients With Acquired Brain Injury as Measured During Physical Activity by POLAR RC810XE Compared to HOLTER EKG
Brief Title: The Reliability of Heart Rate Variability Among Patients With Brain Injury as Measured by POLAR RC810XE Compared to HOLTER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ofer Keren, MD, Sheba Medical Center
Other Study IDs: SHEBA-11-8790-OK-CTIL
Record Dates: First submitted 2011-10-10; First posted 2011-10-13 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Acquired Brain Injury
Keywords: Heart Rate Variability; Acquired Brain Injury; Physical Activity
MeSH Terms: conditions — Brain Injuries; Motor Activity

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- brain injury
  Interventions: Other: no intervention is made

INTERVENTIONS:
Other: no intervention is made — no intervention is made

SUMMARY:
Following a brain injury (BI) in addition to all other systems, there can be a failure in the control of the autonomic system activity. Heart rate (HR) has its own normal variability. Heart rate is controlled by the Sympathetic and Parasympathetic systems. Therefore, monitoring HR variability (HRV) can help us evaluate the balance of the two systems and their efficiency.Decrease in HRV was found to be in correlation with death among patients in the acute stage following ABI. Decrease in HRV is a pre-stage of HR irregularity and ventricular fibrillation.This disturbance can have a great impact on the patients health condition. In addition there was found an inverse correlation between this situation and the rehabilitation outcomes. Based on this data there is a great importance in monitoring HRV during rehabilitation among patients following BI while the patients are required to perform physical activity.The aim of this work is to check whether we can replace the traditional way of measuring HR by EKG Holter (gold standard) with a more simple,accessible tool-the POLAR watch.

The aim of this work is to check if the data collected from a POLAR watch is reliable compared to the data collected from an EKG holter.

ELIGIBILITY:
Inclusion Criteria:

* Brain Injury

Exclusion Criteria:

* a medical condition which doesn't allow the patient to participate physical activity.
* patients that can not be there own legal guardian.
* uncontrolled psychomotoric restlessness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients following brain injury hospitalized in sheba medical center in the Brain injury rehabilitation unit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-10

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Keren, MD, Study Chair — Sheba Medical Center
Locations (1):
- Sheba Medical Center-Brain Injury Rehabilitation Department, Ramat Gan, Israel